CLINICAL TRIAL: NCT00897494
Title: Michigan Center for Pancreatic Cancer Molecular Diagnosis: The Serum Protein Microarray Project
Brief Title: Identification of Biomarkers for Early Detection of Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000479140; P30CA022453 (NIH); WSU-C-2737; WSU-013105MP2E
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Mass Spectrometry; Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: protein expression analysis — Venous blood collection
Other: laboratory biomarker analysis — Venous blood collection
Other: mass spectrometry — Venous blood collection
Other: surface-enhanced laser desorption/ionization-time of flight mass spectrometry — Venous blood collection

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is examining blood samples from patients with cancer to identify biomarkers that may help in the early detection of pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify specific proteins of interest to evaluate for their potential role as markers for pancreatic cancer.
* Analyze serum proteins directly by mass spectrometry to identify new biomarkers of pancreatic cancer that can be used for early diagnosis.

OUTLINE: Blood from patients is collected prior to treatment. Plasma proteins are analyzed by matrix-assisted laser desorption ionization time-of-flight mass spectrometry (MALDI-TOF/MS) and/or electrospray mass spectrometry (ESI/MS).

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of pancreatic cancer

  * Newly diagnosed disease
* Planning to undergo surgery or other treatment for pancreatic cancer at Karmanos Cancer Institute or its affiliates

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Venous blood collection samples from newly dianosed
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2005-02; Primary Completion 2009-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Identification of specific proteins of interest to evaluate for their potential role as markers for pancreatic cancer | Upon collection when patient agrees to provide a one time venous blood collection
Analysis of serum proteins directly by mass spectrometry to identify new biomarkers of pancreatic cancer that can be used for early diagnosis | After separation from the plasma

CONTACTS AND LOCATIONS:
Overall Officials: Fazlul Sarkar, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States